CLINICAL TRIAL: NCT04269811
Title: Phase II Study ofFlu-Bu-Mel Conditioning Regimen for Patients With Myeloid Disease Undergoing Allogeneic Stem Cell Transplantation
Brief Title: Flu-Bu-Mel Conditioning Regimen for Myeloid Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-Myeloid-2020
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Relapse Rate After Allo-HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flu-Bu-Mel (Experimental): Fludarabine 150mg/m2 + Busulfan 3.2mg/kg 2 days + melphalan 50-70mg/m2
  Interventions: Drug: Flu-Bu-Mel

INTERVENTIONS:
Drug: Flu-Bu-Mel — 5-day fludarabine + 2-day busulfan (3.2mg/kg) + 2-day melphalan (50-70mg/m2)

SUMMARY:
For patients with acute myeloid leukemia (AML) or myelodyspasia syndrome undergoing allo-HSCT, the conditioning regimen will be 5-day Fludarabine, 2-day Busulifan and 2-day melphalan

DETAILED DESCRIPTION:
For patients with acute myeloid leukemia (AML) or myelodyspasia syndrome undergoing allo-HSCT, the conditioning regimen will be Fludarabine (30mg/m2, d-7 to d-3) + Busulifan 3.2mg/kg (d-7 to d-6) + melphalan 70mg/m2 (d-4 and d-3). The GVHD prophylaxis will be PT-CY (Cyclophosphamide 50mg/kg d+3 and d+4) + low-dose ATG (2.5mg/kg) on d+15.

ELIGIBILITY:
Inclusion Criteria:

* acute myeloid leukemia (CR1 or CR2) or myelodysplasia syndrome
* patients with HLA matched sibling, unrelated or Haplo-identical donor

Exclusion Criteria:

* patients with active infection
* patients with abnormal liver function damage: ALT/AST above 2X normal range
* patients with abnormal renal function damage Scr>160µmol/L;
* patients with insufficient pulmonary function (FEV1，FVC，DLCO<50%）and heart failure or with EF <50%)
* patients with mental instability or unwilling to give inform consent

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 1 year after transplantation
  From transplantation to documentation of death or relapse or progression

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year after transplantation
  From transplantation to documentation of death due to any causes
Relapse rate | 1 year after transplantation
  From transplantation to documentation of relapse or progression
non-relapse mortality (NRM) | 1 year after transplantation
  From transplantation to documentation of death not due to disease relapse or progression
acute graft versus host disease (aGVHD) | day 180 after transplantation
  Incidence of documented grade II-IV acute GVHD
chronic graft versus host disease (cGVHD) | 1 year after transplantation
  Incidence of documented moderate to severe chronic GVHD
relapse free survival (GRFS) | 1 year after transplantation
  From transplantation to documentation of death, III-IV aGVHD, moderate to severe chronic GVHD and relapse

CONTACTS AND LOCATIONS:
Overall Officials: Jion HU, Principal Investigator — Head BMT program, Rui Jin Hospital
Locations (2):
- China (2):
  - Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai
  - Shanghai No6 Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No